CLINICAL TRIAL: NCT06447506
Title: Long-Term Extension Study (AtDvance) to Evaluate the Safety and Efficacy of GSK1070806 in Participants With Moderate to Severe Atopic Dermatitis.
Brief Title: Long-Term Study (AtDvance) to Evaluate GSK1070806 in Atopic Dermatitis.
Acronym: AtDvance
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor decision to early terminate the study following the termination of the parent study (NCT05999799), which met pre-defined futility criterion for efficacy. No safety concerns were identified.
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 220723; 2023-508474-29-00 (Registry Identifier: CTIS)
Record Dates: First submitted 2024-06-03; First posted 2024-06-07 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Dermatitis, Atopic
Keywords: Atopic dermatits; Dermatitis; Eczema; GSK1070806; Safety; Efficacy; Immune system Disease
MeSH Terms: conditions — Dermatitis, Atopic; Dermatitis; Eczema; Immune System Diseases | interventions — GSK1070806

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: This is a double blinded study until the qualifying parent study has reported out.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- GSK1070806 Dose 1 (Experimental): Participants will receive GSK1070806 Dose 1.
  Interventions: Drug: GSK1070806
- GSK1070806 Dose 2 (Experimental): Participants will receive GSK1070806 Dose 2.
  Interventions: Drug: GSK1070806
- GSK1070806 Dose 3 (Experimental): Participants will receive GSK1070806 Dose 3.
  Interventions: Drug: GSK1070806
- GSK1070806 Dose 4 (Experimental): Participants will receive GSK1070806 Dose 4.
  Interventions: Drug: GSK1070806

INTERVENTIONS:
Drug: GSK1070806 — Participants will receive GSK1070806.

SUMMARY:
The study is designed to evaluate the long-term safety and efficacy of GSK1070806 in participants with moderate-to severe atopic dermatitis, who have completed phase 2b parent GSK atopic dermatitis (AtD) study (NCT05999799).

ELIGIBILITY:
Inclusion Criteria:

* Participants must sign and date the consent document.
* Participants diagnosed with moderate to severe Atopic dermatitis (AtD) who have completed the qualifying Phase 2 parent study (NCT05999799) of GlaxoSmithKline (GSK's) AtD and, in their opinion, may benefit from GSK1070806.
* Be intentional and able to visit the doctor at the clinic by appointment and follow all procedures related to research studies and questionnaires (able to read and understand Patient-reported outcomes (PRO) questionnaires and be able to use electronic devices).
* The use of contraceptive methods for females should be consistent with local regulations on contraceptive methods of participants participating in clinical research programs.
* Female participants are eligible to participate in the research program if they are not pregnant or breastfeeding and meet one of the following conditions:
* It is Woman of nonchildbearing potential (WONCBP).
* It is Woman of childbearing potential (WOCBP) and uses a highly effective contraceptive method that has a failure rate less than (<) 1 percent (%) during the trial dose period and for at least 16 weeks after the last dose of the research drug. We should assess the likelihood of contraceptive failure (e.g., non-cooperation, early contraception) associated with the first dose of the drug.
* WOCBP must obtain a negative result in a highly sensitive pregnancy test (by urine or serum test, as prescribed by local regulations) before receiving the first dose of the research drug.
* If the urine test is positive, or the negative result cannot be confirmed (i.e., the result is unclear), a pregnancy test by serum test is required. In such cases, If the serum is tested, the test result is positive. Participants must be excluded from the research project.
* Additional requirements for testing pregnancy during and after exposure to the drug.
* The researcher is responsible for examining medical history, menstrual cycle history, and sexual activity in the near term. To reduce the risk of screening pregnant women who may not be detected at the beginning of pregnancy.

Exclusion Criteria:

* Permanent discontinuation of the study drug at any time during GSK's qualifying Phase 2 AtD (NCT05999799) or a medical condition that would hinder GSK's participation in the Phase 2 219538 (NCT05999799) AtD research project.
* Participants who, during GSK's qualifying Phase 2 (NCT05999799) AtD research project, developed adverse event (AE) or Serious adverse event (SAE) based on laboratory parameters, physical examination, vital signs, Electrocardiogram (ECG), medical history, etc. Medical history, in the opinion of the researchers, suggests that if Investigational medicinal product (IMP) is continued, it may cause unnecessary risk to the participants.
* Topical medications for AtD within 1 week prior to your appointment at Day 1, such as: Topical calcineurin inhibitors (TCI)/ Topical corticosteroids (TCS), Phosphodiesterase-4 (PDE-4) and Janus activation kinase inhibitors (JAKi) for external use.
* Topical corticosteroids (TCS) (such as hydrocortisone, betamethasone)
* Topical calcineurin inhibitors (TCI) (such as tacrolimus, pimecrolimus)
* Phosphodiesterase-4 (PDE4) inhibitor for external use (e.g., crisaborole)
* JAKi for external use (e.g. ruxolitinib)
* Medications for topical use, or other herbal/traditional medicines that may affect the AtD that the participants are in.
* Participant who received systemic therapy, which is considered contraindicated, including systemic therapy used as a rescue medication for AtD, from the screening for GSK's Phase 2 AtD 219538 research project until the LTE protocol began, were unable to participate in the research project.
* Chronic uncontrolled diseases that may require immediate oral corticosteroids, such as severe uncontrolled asthma (defined as having an Asthma control questionnaire (ACQ)-5 score greater than or equal to (>=) of 1.5 or a history of asthma exacerbations. >= 2 times within the last 12 months, requiring systemic corticosteroid [oral and/or intravenous medication] or requiring a >-24-hour hospital stay)
* Experience participating in previous/current clinical research projects.
* The participants have participated in any other clinical research studies. This is in addition to GSK's Phase 2 219538 (NCT05999799) research project.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2024-06-05 (Actual); Primary Completion 2025-07-29 (Actual); Study Completion 2025-07-29 (Actual)

PRIMARY OUTCOMES:
Number of participants with Adverse event (AE) | Up to Week 280 (End of study [EoS])
  An AE is any untoward medical occurrence in participant, temporally associated with use of study intervention, whether or not considered related to medicinal product.
Number of participants with AE leading to discontinuation of GSK1070806 | Up to Week 280 (EoS)
  An AE leading to discontinuation of GSK1070806 will be reported.
Number of participants with Serious adverse event (SAE) | Up to Week 280 (EoS)
  Any untoward event resulting in death, life threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, congenital anomaly/birth defect, medically important were categorized as SAE.
Number of participants with adverse event of special interest (AESI) | Up to Week 280 (EoS)
  AESI for GSK1070806 include serious infections, opportunistic infections, serious hypersensitivity reactions and injection site reactions (ISRs).

SECONDARY OUTCOMES:
Number of Participants Achieving Investigators Global Assessment (IGA) score of 0 or 1 at Week 16, 32, 48 and up to Week 280 (EoS) | Week 16, 32, 48 and up to Week 280 (EoS)
  IGA for Atopic dermatitis (AtD) is a measure of overall disease severity at the time of assessment on a 5-point scale by the investigator. Where 0-clear, 1-almost clear, 2-mild disease, 3-moderate disease, and 4- severe disease. Higher score indicates severity of disease. A participant with an IGA score of 0 or 1 from baseline will be reported.
Number of participants Achieving Eczema Area and Severity Index (EASI) reduction of greater than or equal to (>=) 75 percent (%) at Week 16, 32, 48 and up to Week 280 (EoS) | Week 16, 32, 48 and up to Week 280 (EoS)
  The occurrence of >=75% reduction from baseline achieving EASI 75 score at Week 16, 32, 48 and up to Week 208 (EoS) will be reported. EASI is an internationally used classification for AtD severity and an investigator-assessed measure that is used to assess the extent (area) and severity of AtD. The range of the scale is 0-72, with a higher score indicating greater severity.
Number of participants with decreased Peak Pruritus Numerical Rating Scale (PP-NRS) by >=4 points at Week 16, 32, 48 and up to Week 280 (EoS) | Week 16, 32, 48 and up to Week 280 (EoS)
  Peak pruritus numerical rating scale (PP-NRS) is a patient reported measure of pruritus (itch) intensity assessing worst itch (in the past 24 hours). The values will be evaluated using an 11-point scale (from 0 to 10), with 0 being no itch and 10 being the worst imaginable itch.
Percentage of participants Achieving maintained response for IGA of 0 to 1 at Week 16, 32, 48 and up to Week 280 (EoS) | Week 16, 32, 48 and up to Week 280 (EoS)
  IGA for AtD is a measure of overall disease severity at the time of assessment on a 5-point scale by the investigator. Where 0-clear, 1-almost clear, 2-mild disease, 3-moderate disease, and 4- severe disease. Higher score indicates severity of disease.
Percentage of participants Achieving maintained response for EASI reduction to >= 75% at Week 16, 32, 48 and up to Week 280 (EoS) | Week 16, 32, 48 and up to Week 280 (EoS)
  The occurrence of >=75% reduction from baseline achieving EASI 75 score at Week 16, 32, 48 and up to Week 208 (EoS) will be reported. EASI is an internationally used classification for AtD severity and an investigator-assessed measure that is used to assess the extent (area) and severity of AtD. The range of the scale is 0-72, with a higher score indicating greater severity.
Percentage change from Baseline in EASI at week 16, 32, 48 and up to Week 280 (EoS) | Week 16, 32, 48 and up to Week 280 (EoS)
  EASI is an investigator-assessed measure that is used to assess the extent (area) and severity of AtD. The range of the scale is 0-72, with a higher score indicating greater severity.

CONTACTS AND LOCATIONS:
Locations (42):
- United States (6):
  - GSK Investigational Site, Fountain Valley, California
  - GSK Investigational Site, Pompano Beach, Florida
  - GSK Investigational Site, Fayetteville, Georgia
  - GSK Investigational Site, New York, New York
  - GSK Investigational Site, Dublin, Ohio
  - GSK Investigational Site, Santa Monica, Texas
- Argentina (4):
  - GSK Investigational Site, Buenos Aires
  - GSK Investigational Site, Ciudad Autonoma de Bueno
  - GSK Investigational Site, Córdoba
  - GSK Investigational Site, Rosario
- Bulgaria (2):
  - GSK Investigational Site, Pleven
  - GSK Investigational Site, Sofia
- Canada (3):
  - GSK Investigational Site, Barrie, Ontario
  - GSK Investigational Site, London, Ontario
  - GSK Investigational Site, Markham, Ontario
- China (3):
  - GSK Investigational Site, Chongqing
  - GSK Investigational Site, Hangzhou
  - GSK Investigational Site, Shanghai
- GSK Investigational Site, Prague, Czechia
- GSK Investigational Site, La Rochelle, France
- Germany (2):
  - GSK Investigational Site, Berlin
  - GSK Investigational Site, Münster
- GSK Investigational Site, Athens, Greece
- Japan (7):
  - GSK Investigational Site, Chiba
  - GSK Investigational Site, Fukuoka
  - GSK Investigational Site, Gunma
  - GSK Investigational Site, Hokkaido
  - GSK Investigational Site, Kanagawa
  - GSK Investigational Site, Osaka
  - GSK Investigational Site, Saitama
- Mexico (3):
  - GSK Investigational Site, Chihuahua City
  - GSK Investigational Site, Durango
  - GSK Investigational Site, Guadalajara
- GSK Investigational Site, Panama City, Panama
- Poland (3):
  - GSK Investigational Site, Elblag
  - GSK Investigational Site, Katowice
  - GSK Investigational Site, Szczecin
- South Korea (2):
  - GSK Investigational Site, Ansan
  - GSK Investigational Site, Seoul
- Spain (3):
  - GSK Investigational Site, Córdoba
  - GSK Investigational Site, Granada
  - GSK Investigational Site, Vigo

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to anonymized individual patient-level data (IPD) and related study documents of the eligible studies via the Data Sharing Portal. Details on GSK's data sharing criteria can be found at: https://www.gsk.com/en-gb/innovation/trials/data-transparency/
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Anonymized IPD will be made available within 6 months of publication of primary, key secondary and safety results for studies in product with approved indication(s) or terminated asset(s) across all indications.
Access Criteria: Anonymized IPD is shared with researchers whose proposals are approved by an Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension may be granted, when justified, for up to 6 months.
URL: https://www.gsk.com/en-gb/innovation/trials/data-transparency/